CLINICAL TRIAL: NCT04067778
Title: A Randomized, Parallel-Group, Non-Inferiority Trial Comparing Random AND Targeted Biopsies to Targeted Biopsies Alone for Neoplasia Screening in Adult Persons With Colonic Inflammatory Bowel Diseases: A Pilot Study
Brief Title: IBD Neoplasia Surveillance Pilot RCT
Acronym: IBDDysplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Health Sciences Centre, Winnipeg, Manitoba (Other); Western University, Canada (Other); University of Toronto (Other); Hamilton Health Sciences Corporation (Other); Thunder Bay Regional Health Sciences Centre (Other); Eastern Health (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Providence Health & Services (Other); Royal Jubilee Hospital (Unknown); University of Alberta (Other); MOUNT SINAI HOSPITAL (Other); Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20190428-01T
Record Dates: First submitted 2019-08-07; First posted 2019-08-26 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Inflammatory Bowel Diseases; Colonic Neoplasms; Dysplasia
Keywords: IBD; Dysplasia; Biopsy; Colonoscopy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will undergo standard colonoscopy as part of their routine IBD surveillance. During this colonoscopy targeted biopsies (biopsies of any pre-cancerous lesions observed by the doctor) and/or removal of any polyps will be undertaken.
  Interventions: Diagnostic Test: Intervention Group
- Control Group (Other): Participants will undergo standard colonoscopy as part of their routine IBD surveillance. During this colonoscopy both random (approximately 32 to 40) and targeted biopsies (and/or removal of any polyps) will be undertaken.
  Interventions: Diagnostic Test: Control Group

INTERVENTIONS:
Diagnostic Test: Intervention Group — Standard colonoscopy with targeted biopsies only
  Arms: Intervention Group
Diagnostic Test: Control Group — Standard colonoscopy with random AND targeted biopsies
  Arms: Control Group

SUMMARY:
To determine if random biopsies can be safely eliminated from screening of average risk persons with IBD, the investigators propose to carry out a pilot randomized control trial in which targeted biopsies in combination with random biopsies will be compared to targeted biopsies alone in terms of pre-cancerous lesion capture rate, side-effects and CRC risk. The pilot study will aim to capture 20% of the overall study population in order to evaluate the feasibility of recruiting the needed number of participants in the specified time frame, while maintaining high quality of data collection.

DETAILED DESCRIPTION:
Inflammatory Bowel Disease (IBD), including crohn's disease and ulcerative colitis, is a group of diseases characterized by acute and chronic inflammation of the intestinal tract. Persons with IBD are at an increased risk of developing colorectal cancer (CRC) and require frequent CRC screening with colonoscopy. Current IBD screening guidelines recommend the taking of biopsies of any lesions suspected to be pre-cancerous (targeted biopsies), as well as the taking of 30 to 40 random biopsies throughout the colon. The recommendations for random biopsies are based on historical practice and the theory that they would capture "invisible lesions", but are not supported by strong scientific evidence.

In fact, recent evidence has shown that random biopsies capture a very small number of pre-cancerous lesions and that they capture such lesions only in persons with additional risk factors for CRC. In addition, new colonoscopy practices and technology have made 80-90% of pre-cancerous lesions visible. Random biopsies also carry potential risks for patients, including lower gastrointestinal bleeding and bowel perforation, and substantially increase procedural costs and time.

Hence, there is a strong impetus to conduct a well-powered non-inferiority Randomized Controlled Trial (RCT) on this topic in a Canadian setting. With the support of a pan-Canadian IBD clinical trials alliance (the Canadian IBD Research Consortium (CIRC)), and the high prevalence of IBD in Canada, Canadian investigators are well-positioned to undertake such a trial. Before embarking on a large multi-center trial, a one-year pilot feasibility trial will be conducted to ensure that patients can be enrolled efficiently with excellent protocol compliance. A feasibility trial will also provide a crude estimate of the neoplasia detection rate (primary outcome) among persons with colon IBD (cIBD) in Canada, which will allow refinement of the sample size, recruitment period and budget for a definitive trial. To-date, no well-powered or North American RCTs have evaluated random biopsies as an intervention to guide our estimates for a definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Historical endoscopic/histologic disease extending beyond the rectum in UC or involving ≥ 1/3 of colorectum in CD
* > 50% of colon present, with remaining colon meeting above minimum criteria for disease extent (beyond rectum in UC, ≥1/3 colorectum in CD
* cIBD ≥ 8 years duration (or at any time after diagnosis if a patient also has primary sclerosing cholangitis)
* In symptomatic remission at time of colonoscopy

  * For CD: Harvey-Bradshaw Index < 541
  * For UC or IBDU: Partial Mayo Score ≤ 242
* Major purpose of colonoscopy is neoplasia screening/surveillance
* Undergoing colonoscopy with high-definition white light endoscopy

Exclusion Criteria:

* Persons who cannot or are unwilling to provide informed consent
* Persons with a history of colorectal cancer
* Persons with prior subtotal or total colectomy (> 50% of colon removed)
* Persons undergoing colonoscopy to follow-up on recently diagnosed neoplasia identified within the past year
* Persons undergoing pancolonic chromoendoscopy
* Colon mucosa visibility deemed inadequate for surveillance after washing/suctioning (Boston Bowel Preparation Score of 0 or 1 in any segment)
* Incomplete colonoscopy (unable to reach cecum)
* Moderate-to-severe inflammation (Mayo 2-3) involving ≥ 25% of colorectum or mild inflammation (Mayo 1) involving ≥ 50% of colorectum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Overall Number of Participants Enrolled | 1 year
  Number of participants enrolled within one year from the overall total required.
Rate of Protocol Adherence | 1 year
  Rate of protocol adherence of major protocol violations on a per-patient basis.
Rate of overall neoplasia detection | 1 year
  Overall neoplasia detection rate for the definitive trial.
Adverse Events occurrence | 2 weeks
  Occurrence of serious and minor post-procedural adverse events within 2 weeks of procedure.

SECONDARY OUTCOMES:
Rate of Study Variables | 1 year
Rate of Missed 2-Week Post-Procedural Assessment for Complications | 2 weeks

CONTACTS AND LOCATIONS:
Locations (12):
- Canada (12):
  - University of Alberta, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Pacific Digestive Health / Royal Jubilee Hospital, Victoria, British Columbia
  - University of Manitoba, Health Sciences Centre, Winnipeg, Manitoba
  - Eastern Regional Health Authority, St. John's, NFLD
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - London Health Sciences Centre, University Hospital, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Derived] Murthy SK, Marderfeld L, Fergusson D, Ramsay T, Bernstein CN, Nguyen GC, Jairath V, Riddell R. A randomized trial evaluating the utility of non-targeted biopsies for colorectal neoplasia detection in adults with inflammatory bowel disease: a pilot study protocol. Pilot Feasibility Stud. 2024 Feb 1;10(1):20. doi: 10.1186/s40814-023-01434-8. PMID 38297397